CLINICAL TRIAL: NCT01148563
Title: LSU HCSD Tele-Health Projects: Adult Systolic Heart Failure Patient Population
Brief Title: Louisiana State University Health Care Sciences Division (LSU HSCD) Tele-Health Projects: Adult CHF Patient Population
Acronym: TeleHealth:CHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PBRC 29003
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Congestive Heart Failure
Keywords: congestive heart failure; systolic; chronic disease; heart failure
MeSH Terms: conditions — Heart Failure; Systolic Murmurs; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (No Intervention): The Standard Care group will continue regular LSU HCSD disease management care for heart failure patients with no additional intervention.
- Tele-health Monitoring Group (Active Comparator): The tele-monitoring intervention group will have the continual standard care from their physician plus the tele-health monitoring. The tele-health monitor will collect the following data: weight, blood pressure, pulse oximetry, pulse rate, & patient responses to disease-specific questions regarding changes in state of health for 6 months.
  Interventions: Device: Tele-health Monitoring

INTERVENTIONS:
Device: Tele-health Monitoring — Daily tele-health monitoring data will be collected from randomized participants.
  Arms: Tele-health Monitoring Group

SUMMARY:
The purpose of this research study is to see whether a tele-health intervention can improve health, functioning status, emotional status, quality of life, and patient satisfaction for patients with Congestive Heart Failure (CHF) and to examine the cost benefits of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* equal to or greater than 18 years old
* 1 + past CHF diagnosis in LSU database, with history of CHF diagnosis extending back for 12 months
* LSU primary care or chronic disease clinic patient for equal or greater than 6 months.
* On CHF medication for equal to or greater than 6 months
* Have had a past echocardiogram
* Mental competency to consent and participate (determined by clinical judgment and chart abstraction)
* Physically able to use in-home equipment (or presence of a household member who can assist the subject in equipment use)
* Currently-working conventional telephone line at primary residence
* Grounded electrical power supply at primary residence
* Anticipation of remaining in the LSU HCSD patient population for the next year
* Not on home oxygen therapy
* No planned surgery within the next six months
* Living at home (not institutionalized)
* No history of major organ transplant
* No diagnosis of metastatic or inoperable cancer
* Not under treatment for cancer
* Not under treatment for end-stage renal disease or end-stage liver disease
* 1 + emergency department visit or inpatient stay in past 12 months

Exclusion Criteria:

* Are on home oxygen
* Have a planned surgery within the next 6 months
* Have a history of major organ transplant
* Have a diagnosis of metastatic or inoperable cancer
* Are under treatment for cancer
* Are under treatment for end-stage renal disease or end-stage liver disease
* Have HIV/AIDS
* Have a cognitive condition, such as Alzheimer's or dementia that would make it difficult for you to understand how to use the tele-health device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Arcement, MD, Principal Investigator — Louisiana State University Health Care Services Division; Michael Kaiser, MD, Study Chair — Louisiana State University Health Care Services Division; Ronald Horswell, PhD, Study Chair — Louisiana State University Health Care Services Division; Jay Besse, BS, Study Chair — Louisiana State University Health Care Services Divison; Timothy S. Church, MD, MPH, PhD, Study Chair — Pennington Biomedical Research Center; Valerie H. Myers, PhD, Study Chair — Pennington Biomedical Research Center; Donna H. Ryan, MD, Study Chair — Pennington Biomedical Research Center
Locations (4):
- United States (4):
  - Earl K. Long Medical Center, Baton Rouge, Louisiana
  - Leonard J. Chabert Medical Center, Houma, Louisiana
  - University Medical Center, Lafayette, Louisiana
  - WO Moss Regional Medical Center, Lake Charles, Louisiana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were nested within LSU HCSD clinics. Potential subjects were approved by their physicians for inclusion in addition to meeting the stated inclusion criteria.
  Study recruiters contacted the potentially-eligible subjects at the times of their next scheduled clinic visits. Recruitment Period: 3/9/09-8/31/10.
Pre-assignment Details: Of the original 137 subjects recruited, one subject in the treatment group withdrew from the study prior to having home monitoring equipment installed, leaving a total of 136 subjects.
Period: Overall Study
Arm/Group | Standard Care | Tele-health Monitoring Group
Started | 69 | 67
Completed | 40 | 37
Not Completed | 29 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Tele-health Monitoring Group | Total
Number analyzed (Participants) | 69 | 67 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 54 | 106
  >=65 years | 17 | 13 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.623188 (9.2801202) | 56.641791 (10.08855) | 57.139706 (9.6633502)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 29 | 69
  Male | 29 | 38 | 67
Region of Enrollment [Number; unit: participants]
  United States | 69 | 67 | 136

OUTCOME MEASURES:

1. Primary Outcome: Events Per Person-year
Description: (Number of emergency department visits + number of inpatient stays) / person-year
Time Frame: 12 months
Population: Used an Intention to Treat (ITT) Analysis. Missing outcome data were imputed as necessary.
Measure: Mean (95% Confidence Interval); unit: events/person-year
Arm/Group | Standard Care | Tele-health Monitoring Group
Number analyzed (Participants) | 69 | 67
events/person-year | 84 [66 to 106] | 57 [43 to 76]
Statistical Analysis 1: Comparison: Standard Care vs Tele-health Monitoring Group; Test type: Superiority; p = 0.094, bootstrapping; Risk Ratio, log = -0.30, 95% CI 2-sided [-0.65 to 0.05], Standard Error of Mean 0.18 — The hypothesis test was based on ln(relative risk), with the tele-monitoring group value as the relative risk numerator and the control group value as the denominator. The standard error was generated by bootstrapping the sample

2. Secondary Outcome: U.S. Dollars Per Person-year
Description: (emergency department costs + inpatient costs) / person-year
Time Frame: 12 months
Population: All heart failure patients included in the study
Measure: Mean (Standard Error); unit: U.S. dollars per person-year
Arm/Group | Standard Care | Tele-health Monitoring Group
Number analyzed (Participants) | 69 | 67
U.S. dollars per person-year | 10363 (1630) | 7212 (279)
Statistical Analysis 1: Comparison: Standard Care vs Tele-health Monitoring Group; Test type: Superiority; p = 0.105, bootstrapping; The standard error was generated by bootstrapping the sample; Risk Ratio, log = .70, 95% CI 2-sided [0.45 to 1.08], Standard Error of Mean 0.22 — The hypothesis test was based on ln(relative risk) with the tele-monitoring group value as the numerator and the control group as the denominator

ADVERSE EVENTS:
Time Frame: 6 months per participant
Description: The adverse events were identified via both care management interaction with patients and by electronic medical record data.
Arm/Group | Standard Care | Tele-health Monitoring Group
Serious Adverse Events (participants affected / at risk) | 40/69 | 31/67
Other Adverse Events (participants affected / at risk) | 0/69 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=69) | Tele-health Monitoring Group (N=67)
Any ER visit or Inpatient stay (General disorders) | 40 (86) | 31 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No